CLINICAL TRIAL: NCT00236925
Title: A Double-Blind Crossover Within Subject Study on Low-Dose Hydrocortisone for Fibromyalgia
Brief Title: Efficacy Study of Low-Dose Hydrocortisone Treatment for Fibromyalgia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Gustav Schelling,MD, Senior Researcher, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 348/02
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Cortisol; Hydrocortisone; Stress
MeSH Terms: conditions — Fibromyalgia | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose Hydrocortisone (Active Comparator): Low Dose Hydrocortisone
  Interventions: Drug: Low dose Hydrocortisone; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Low dose Hydrocortisone; Drug: Placebo

INTERVENTIONS:
Drug: Low dose Hydrocortisone — Hydrocortisone 10 mg daily
  Other Names: Cortisol
Drug: Placebo — Placebo

SUMMARY:
This study is based on clinical findings that some patients with fibromyalgia have a tendency towards lower levels of the stress hormone cortisol. The hypothesis to be tested in this study is that the administration of a very low-dose of cortisol which has no side effects corrects this deficiency and results in an improvement of symptoms

DETAILED DESCRIPTION:
Fibromyalgia (FMS) is regarded as one of the most important chronic pain syndromes with a high prevalence in the general population.

Hypotheses to be tested in this study:

* Impaired glucocorticoid signaling is associated in a failure to terminate the chronic stress response seen in patients with FMS.
* Low-dose hydrocortisone in patients with FMS results in a reduction in pain and other stress-related symptoms of FMS

Intervention:

2 x 5 mg of hydrocortisone given at noon and in the evening

Study design:

Double-blind, randomized, cross-over, within-subject

Presumed mechanism of main hydrocortisone effect:

* Improvements in FMS symptoms representing (functional) hypocortisolism
* Increased pain threshold

Expected results:

* Moderate reductions in physical impairment, fatigue, and stiffness
* Improvements in sleep quality
* Decline in pain intensity Inclusion criteria
* FMS diagnosis according to the American College of Rheumatology 1990 Criteria
* Age between 18 and 60 years

Exclusion criteria

* Disease states representing contraindications to the administration of glucocorticoids (tuberculosis, gastric- and duodenal ulcers, Cushing's disease, osteoporosis, hypertension, pregnancy and lactation, psychosis, glaucoma, diabetes mellitus, thrombophilia, active or chronic bacterial or viral infections, hypothyreosis, cirrhosis).
* Severe or chronic somatic diseases.
* Psychiatric diseases according to DSM-IV (except PTSD, minor depressive episodes, minor personality disorders).
* Body weight >20% above or below normal.
* Changes in pharmacologic or psychotherapeutic management less than 3 months ago.
* Age < 18 years

Proposed outcome measures

* Primary: FMS symptoms, pain scores, tenderness at tender points
* Secondary: Chronic stress symptoms, health-related quality of life

Possible benefit and use of data from the trial

This trial could help to identify glucocorticoid resistance as a major mechanism underlying the sustained stress - reactions seen in FMS and establish low-dose hydrocortisone as a useful drug for treatment of stress-related disorders.

ELIGIBILITY:
Inclusion Criteria:

* FMS diagnosis according to the American College of Rheumatology 1990 Criteria.
* Age between 18 and 60 years

Exclusion Criteria:

* Disease states representing contraindications to the administration of glucocorticoids (tuberculosis, gastric- and duodenal ulcers, Cushing's disease, osteoporosis, hypertension, pregnancy and lactation, psychosis, glaucoma, diabetes mellitus, thrombophilia, active or chronic bacterial or viral infections, hypothyreosis, cirrhosis)
* Severe or chronic somatic diseases
* Psychiatric diseases according to DSM-IV (except PTSD, minor depressive episodes, minor personality disorders)
* Body weight >20% above or below normal
* Changes in pharmacologic or psychotherapeutic management less than 3 months ago
* Age < 18 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-05; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia symptoms | 3 months

SECONDARY OUTCOMES:
Chronic stress symptoms | 3 months
Health-related quality of life | 3 months
Life satisfaction | 3 months
Infection | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Schelling, MD, PhD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Ludwig-Maximilians University, Munich, Bavaria, Germany

REFERENCES:
- [Background] Aerni A, Traber R, Hock C, Roozendaal B, Schelling G, Papassotiropoulos A, Nitsch RM, Schnyder U, de Quervain DJ. Low-dose cortisol for symptoms of posttraumatic stress disorder. Am J Psychiatry. 2004 Aug;161(8):1488-90. doi: 10.1176/appi.ajp.161.8.1488. PMID 15285979
- See also: Homepage of the Dept. of Anaesthesiology of the University of Munich — http://ana.klinikum.uni-muenchen.de/